CLINICAL TRIAL: NCT02920827
Title: A Double-Blind, Randomised, Placebo-Controlled Safety and Pharmacokinetic Trial in Healthy HIV-Negative Women to Assess Delivery of Dapivirine From the Matrix Vaginal Ring Containing 25 MG of Dapivirine
Brief Title: Safety and Pharmacokinetic Trial in Healthy HIV-Negative Women to Assess the Delivery of Dapivirine From a Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM024; NCT01144013 (obsolete NCT alias)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections
Keywords: HIV Infections; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapivirine Vaginal Ring (Experimental): Vaginal ring containing 25 mg dapivirine
  Interventions: Combination Product: Dapivirine Vaginal Ring
- Placebo Vaginal Ring (Placebo Comparator): Placebo vaginal ring
  Interventions: Combination Product: Placebo vaginal ring

INTERVENTIONS:
Combination Product: Dapivirine Vaginal Ring — A platinum-catalysed silicone elastomer matrix vaginal ring containing 25mg of dapivirine used over 28 days
  Arms: Dapivirine Vaginal Ring
Combination Product: Placebo vaginal ring — Placebo vaginal ring containing no dapivirine
  Arms: Placebo Vaginal Ring

SUMMARY:
The proposed study is a single center, double-blind placebo-controlled trial to assess the safety and tolerability of the dapivirine ring as compared to a placebo ring when inserted for 28 days in 16 healthy, HIV-negative women.

DETAILED DESCRIPTION:
The objective of this trial was to evaluate the feasibility of using a platinum-catalyzed matrix vaginal ring, containing 25 mg of dapivirine, to deliver investigational product for 28 continuous days. The specific objectives were to:

1. Assess the safety and tolerability of the vaginal ring containing dapivirine, when used continuously for 28 days, compared to a placebo ring
2. Assess dapivirine concentrations in plasma before, during and after 28 days' use of a silicone elastomer matrix vaginal ring containing dapivirine
3. Assess dapivirine concentrations in vaginal fluids before, during and after 28 days' use of a silicone elastomer matrix vaginal ring containing dapivirine. Safety was evaluated from clinical evaluations, clinical laboratory test results and adverse events (AEs). The pharmacokinetic (PK) evaluation was made based on systemic absorption from plasma concentrations and local disposition from vaginal fluid concentrations.

ELIGIBILITY:
Inclusion Criteria:

* were females between 18 and 40 years of age, inclusive
* were willing and able to give written, informed consent
* were available for all visits and consented to follow all procedures scheduled for the trial
* were healthy, based on medical history, vital signs, physical examination, urinalysis (dipstick and microscopy), laboratory evaluations for genital infections (gonorrhea, chlamydia and trichomonas), and laboratory evaluations for hematology and biochemistry
* were HIV-negative, as determined by an HIV test at screening
* were willing to abstain from sexual activity for the duration of the period of ring use
* were on a stable form of contraception, defined as a stable oral contraceptive regimen for at least two months prior to enrollment; OR a transdermal contraceptive patch for at least three months prior to enrollment; OR long-acting progestins for at least six months prior to enrollment; OR had an intra-uterine device (IUD) inserted (with no vaginal or gynecological complaints associated with its use) at least three months prior to enrollment; OR had undergone surgical sterilization at least three months prior to enrollment; AND were willing to use oral contraceptives, if necessary, to avoid menstruation while taking part in this trial
* were asymptomatic for genital infections at the time of enrollment, and the cervix and vagina appeared normal upon pelvic examination and colposcopy, as determined by the investigator
* were willing to refrain from the use of vaginal products or objects including, but not limited to, tampons, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, non-trial vaginal rings and drying agents for 14 days prior to enrollment and for the duration of the trial
* were willing to refrain from participation in any other research trial for the duration of this trial
* were willing to provide adequate locator information for trial retention purposes and were reachable per local standard procedures (e.g. by home visit or telephone, or via family or close neighbor contacts (confidentiality was to be maintained))
* were hepatitis B and C negative at the time of screening.

Exclusion Criteria:

* had a history of anaphylaxis or severe allergy resulting in angioedema, or a history of sensitivity/allergy to latex or silicone
* were pregnant or breast-feeding, or had their last pregnancy outcome within three months prior to screening
* were participating in any other clinical research trial involving investigational or marketed products at the time of this trial or within two months prior to screening
* had a history or diagnosis of and/or treatment for a sexually transmitted disease within the previous three months
* had a history of genital tract surgery within the previous two months
* had a current diagnosis of sexually transmitted infections (STIs) (gonorrhea, chlamydia and/or trichomonas)
* had current vulvar or vaginal symptoms/abnormalities that could influence the trial results
* had a history of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding or urethral obstruction, incontinence or urge incontinence
* had symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection
* had current non-iatrogenic pelvic/colposcopic examination findings involving deep epithelial disruption
* had any Grade 2, 3 or 4 hematology, biochemistry or urinalysis laboratory abnormality at baseline (screening), according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading Adverse Events
* had a Pap test result at screening that required cryotherapy, biopsy, treatment (other than for infection) or further evaluation; this included any findings of atypical squamous cells of undetermined significance (ASCUS)
* had any condition(s) that, in the opinion of the investigator, could interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety: To assess the safety and tolerability of the dapivirine vaginal ring, the endpoint was the proportion of women on the dapivirine or placebo ring experiencing specific, protocol-defined safety events during the study (see description). | 28 days
  * mucosal abnormalities (as defined in the CONRAD/WHO manual) visible during naked eye examination and/or colposcopy
  * positive diagnostic tests for trichomonas, gonorrhea, and/or chlamydia
  * at least one AE during the trial period
  * any laboratory abnormalities on hematology and biochemistry
  * abnormal vaginal pH and/or abnormal vaginal flora during the course of the trial.
Pharmacokinetics: assessed by measurement of the concentrations of dapivirine in plasma and in vaginal fluids (collected by Tear Test Strips) before, during and after the trial period. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Annalene Nel, PhD, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (1):
- SGS Life Sciences Center, Antwerp, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided